CLINICAL TRIAL: NCT00511615
Title: A Feasibility Study of Molecular Imaging for Detection of Cervical Intraepithelial Neoplasia
Brief Title: Molecular Imaging for Detection of Cervical Intraepithelial Neoplasia
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2004-0862
Record Dates: First submitted 2007-08-02; First posted 2007-08-06 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Cervical Cancer
Keywords: Cervical Intraepithelial Neoplasia; Loop Electrosurgical Excision Procedure; Cervical Cancer; Colposcopy; Molecular Imaging; LEEP
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue sample removal from the cervix using LEEP during the scheduled colposcopy.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with cervical cancer scheduled to be treated with the LEEP procedure.
  Interventions: Procedure: Loop Electrosurgical Excision Procedure (LEEP)

INTERVENTIONS:
Procedure: Loop Electrosurgical Excision Procedure (LEEP) — Tissue sample removed from cervix using LEEP and contrast agent.
  Other Names: LEEP

SUMMARY:
The hypothesis of this research project is that topical application of the anti-EGFR or anti-E6/E7 contrast agents followed by optical imaging will yield images that reflect spatial variations in expression that correlate with the presence of cervical precancer. To gather feasibility data the investigators will:

1. Obtain cervical specimens from women with high grade squamous intraepithelial lesions (HGSILs) being treated with the loop electrosurgical excision procedure (LEEP).
2. After Loop Electrosurgical Excision Procedure (LEEP) is performed, obtain low and high resolution optical images before and after applying contrast agents topically to the epithelial surface of the tissue for 30 minutes before rinsing.
3. Submit the specimen for histology, and have it sectioned and stained using both H&E and immunohistochemical staining for EGFR or E6/E7. The images will be reconstructed into a two dimensional map delineating areas of Cervical Intraepithelial Neoplasia (CIN) and of EGFR or E6/E7 overexpression. Maps of the pathology will be compared to those obtained from the intact cervix exposed to the contrast agent.

DETAILED DESCRIPTION:
During your scheduled colposcopy, a sample of tissue will be removed from your cervix using the loop electrosurgical excision procedure (LEEP). The LEEP is the standard of care treatment for the precancerous condition on your cervix. The details of the procedure will be covered in another consent form. Before the LEEP, a photograph will be taken of the cervix. This photograph will be taken for research purposes, so that researchers will have a photograph to compare to the images taken with the MDC and Confocal.

The tissue that is removed will be taken to a room where the researchers will use a special microscope to look at the tissue before and after the new contrast agent is painted on the surface of the tissue. After the tissue samples are looked at, they will be sent to the lab for routine tests (as part of your standard of care).

You will require a LEEP whether you participate in this study or not. The tissue removal is a standard part of the LEEP. The experimental portion of this study is the use of the contrast agent. Once that portion is complete, the tissue will be tested as per standard of care. The tissue will not be used for any other research testing.

You will not be told of any of the experimental findings with the contrast agent. However, your doctor and/or nurse practitioner will be told the results of the routine tests, and they will give these results to you.

This is an investigational study. The LEEP is considered standard of care and any charges associated with the LEEP will be the responsibility of you and/or your insurance provider. Up to 80 women will take part in this multicenter study. Up to 40 will be enrolled at M.D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are 18 years of age or older.
2. Patients who are not pregnant.
3. Patients who are not HIV positive.
4. Patients who are scheduled to be treated for SIL with LEEP.

Exclusion Criteria:

1. Patients who are younger than 18 years of age.
2. Patients who are pregnant.
3. Patients who are HIV positive.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cervical cancer scheduled to be treated with the LEEP procedure.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2005-03; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To learn if a new type of contrast agent (a dye used in certain types of scans and microscope studies) can be used to detect cervical cancer and precancerous lesions better than standard contrast agents. | 4 Years

CONTACTS AND LOCATIONS:
Overall Officials: Michele Follen, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (3):
  - Lyndon B. Johnson Hospital, Houston, Texas
  - U.T.M.D. Anderson Cancer Center, Houston, Texas
  - UT Health Science Center-Houston, Houston, Texas
- British Columbia Cancer Agency, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Aaron J, Nitin N, Travis K, Kumar S, Collier T, Park SY, Jose-Yacaman M, Coghlan L, Follen M, Richards-Kortum R, Sokolov K. Plasmon resonance coupling of metal nanoparticles for molecular imaging of carcinogenesis in vivo. J Biomed Opt. 2007 May-Jun;12(3):034007. doi: 10.1117/1.2737351. PMID 17614715
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org